CLINICAL TRIAL: NCT02933047
Title: Laparoscopic Hysterectomy - A Randomized Controlled Trial on Outpatient Versus Inpatient Regimen
Brief Title: Laparoscopic Hysterectomy - Outpatient Versus Inpatient Regimen
Acronym: LH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5711674; 1-16-02-212-13 (Other: Danish Dataprotection Agency)
Record Dates: First submitted 2013-10-21; First posted 2016-10-14 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2016-04

CONDITIONS: Outpatient Hysterectomy
Keywords: Hysterectomy; Patient satisfaction; Rehabilitation; Laparoscopy; Return to work; Exercise
MeSH Terms: conditions — Patient Satisfaction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outpatient LH (Active Comparator): Patients in the intervention group are discharged within 6 to 8 hours after total laparoscopic hysterectomy.
  Interventions: Procedure: Total laparoscopic hysterectomy
- Inpatient LH (Placebo Comparator): Patients in the control group follow regular hospitalization and are discharged within 24 hours after total laparoscopic hysterectomy.
  Interventions: Procedure: Total laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Total laparoscopic hysterectomy
  Arms: Outpatient LH
Procedure: Total laparoscopic hysterectomy
  Arms: Inpatient LH

SUMMARY:
Laparoscopic Hysterectomy (LH) is increasingly used as a standard surgical approach to hysterectomy. It is a safe procedure with low rates of complications and readmissions. Increasing evidence indicates that LH may be suitable for an outpatient setting but this may impair patient's satisfaction in more than 25% of cases. In addition, change from in-patient care to day case surgery might influence readmission rates and postoperative physical activity. No data are available on the current length of sick leave in Danish patients after hysterectomy, and the effects of outpatient surgery on this parameter are difficult to predict. A randomized controlled trial of LH performed as an outpatient procedure compared with today's inpatient standard will provide a firm platform for future planning of routine treatment of patients with need of hysterectomy for benign indications.

DETAILED DESCRIPTION:
Hysterectomy is the most frequent gynecological operation world wide and the indication is often benign. The women are healthy and young with a median age below 50 years. In Denmark, hysterectomy is performed as an inpatient procedure with a median hospitalization of 1 day. Hysterectomies in Denmark are distributed by 45% abdominal hysterectomies (AH), 35% vaginal hysterectomies (VH) and 20% laparoscopic hysterectomies (LH). There is no final consensus whether VH or LH should be recommended as first choice but LH is gaining more and more acceptance. Increasing evidence indicates that LH may be suitable for an outpatient setting. Data seem to assure that outpatient LH is feasible but patient's satisfaction in this setting remains an open question. A detailed analysis of data from a Norwegian study indicates that patients reporting dissatisfaction with the early discharge amounts to 25-38%. Such a decrease in patient's satisfaction would present a significant problem, and a randomized controlled study of sufficient size with focus on this aspect is therefore needed.

Recommendations on postoperative sick leave vary considerably, due to lack of evidence-based guidelines and no firm data are available on the relation between outpatient treatment and sick leave in gynecology.

This randomized controlled study attempt to examine outpatient LH and patient satisfaction and related subject as readmissions and complications, time to return to work, physical activity in the recuperation period and an overall socioeconomic calculation of the costs of LH in an in- and outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women below 56 years who is in need of a hysterectomy for benign conditions.
* Additional surgery is allowed in the gynecological area.
* BMI and working status is NOT exclusion criteria's.

Exclusion Criteria:

* Unable to read and write Danish to answer questionnaires.
* Unable to walk to carry a pedometer.

Ages: 18 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Satisfaction with length of stay after total laparoscopic hysterectomy. | 2 weeks after surgery
  Difference in satisfaction with length of stay between intervention group and placebo measured on a visual analogue scale from 0 to 10 with 10 being most satisfied and presented on an international unit scale.
Patient satisfaction and quality of life | 4 weeks from date of surgery
  The difference in patient satisfaction between inpatient and outpatient laparoscopic hysterectomy 4 weeks from surgery measured by the European Quality of life questionnaire in 5 dimensions (EQ5D) and presented as an index number.

SECONDARY OUTCOMES:
Incidence and pattern of complications and readmissions for in- and outpatient LH. | 4 weeks from the date of surgery
  Number and type of complications found in medical records. Outcome will be presented as odds ratios and compared using chi2 measurement.
Physical activity in the recovery period after in- and outpatient LH. | 4 weeks from the date of surgery
  Daily walking distance in steps per day. Data will be presented as repeated measurement and the groups are compared by pairwise comparison.
Return to work after in- and outpatient LH. | 6 month from the date of surgery
  Date of return to work after surgery. The sick-leave is 14 days. When the sick-leave is more than 14 days it will be part of a socioeconomic analysis of lost work capacity and time spend on consultations. The difference between the groups will be measured in QALY's (Quality adjusted life year) and monetary values.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla J. Christiansen, MD, Principal Investigator — Arhus University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christiansen UJ, Kruse AR, Olesen PG, Lauszus FF, Kesmodel US, Forman A. Outpatient vs inpatient total laparoscopic hysterectomy: A randomized controlled trial. Acta Obstet Gynecol Scand. 2019 Nov;98(11):1420-1428. doi: 10.1111/aogs.13670. Epub 2019 Jul 15. PMID 31148146